CLINICAL TRIAL: NCT01389570
Title: Postoperative Nausea/Vomiting and Acupressure Can Acupressure With Wristbands Reduce the Use of Antiemetics for the Treatment of Postoperative Nausea and Vomiting?
Brief Title: Postoperative Nausea/Vomiting and Acupressure
Acronym: Acunausea
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Research Centre of Complementary and Alternative Medicine, Norway (Other)
Collaborators: Lovisenberg Diakonale Hospital (Other)
Responsible Party: Arne Johan Norheim, National Research Centre of Complementary and Alternative Medicine, Norway
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011/176
Record Dates: First submitted 2011-05-31; First posted 2011-07-08 (Estimated); Last update posted 2011-07-18 (Estimated); Status verified 2011-06

CONDITIONS: Postoperative Nausea
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acupressure wrist band (Experimental): The group receiving acupressure wrist band
  Interventions: Procedure: Acupressure wrist band

INTERVENTIONS:
Procedure: Acupressure wrist band — Use of acupressure wristband during surgery Manufacturer; Pinnacle Ind Ltd, Rm 831 Thriving Ind Ctr, 26-38 Sha Tsui Rd, Tsuen Wan, Hong Kong
  Other Names: Sea-Band Ltd

SUMMARY:
Postoperative nausea and vomiting (PONV) remain a significant challenge in our practice. However, pharmaceutical prophylaxis can confer unpleasant adverse effects. It would therefore be appropriate to consider the use of non-pharmacological methods in preventing PONV. Acupuncture and acupressure are reported to be effective preventive treatment for PONV, and the adverse effects are minimal. Consequently, the aim of the study is to implement acupressure in our anaesthetic department procedures. A reduction of the use of antiemetics will be a parameter on the effectiveness of acupressure. The study will focus on acupressure as a supplement to the ordinary prophylactic treatment of PONV in adults undergoing orthopaedic and general surgery, and adults and children undergoing ear, nose, throat surgery. The primary endpoints are the quantities of antiemetics used before (baseline) and during the implementation period. The study will be conducted from January to December 2011.

DETAILED DESCRIPTION:
Background:

Nausea and vomiting after surgery and anaesthesia are inconvenient and undesirable physiological and psychological events. In addition to causing distress and discomfort for the patient, retching and vomiting can increase the risk of pain and bleeding, resultant resource use, and prolong stay at the postoperative ward and hospital. The mechanisms behind Postoperative nausea and vomiting (PONV) are complicated, and many of the trigger factors are still unknown. Several types of pharmaceutical antiemetics are in use, but drug therapy is only partially effective in preventing or treating PONV. In 2008 we conducted a trial to assess the effectiveness of acupuncture and acupressure (acustimulation) in reducing postoperative retching and vomiting in children undergoing tonsillectomy and/or adenoidectomy. The results were promising, and the article is published in Acupuncture in Medicine in March 2011.

Acustimulation:

Cochrane systematic reviews show the effect of acupuncture and acupressure in postoperative antiemetic treatment. The reviews show no clear difference in the effectiveness of P6 acupoint stimulation for adults and children, or for invasive and non-invasive acupoint stimulation. Moreover, there was no reliable evidence for differences in risks of postoperative nausea or vomiting after P6 acupoint stimulation compared to antiemetic drugs.

Aim and objective:

Acupressure wrist bands are less expensive compared to most antiemetics, and the adverse effects of acupoint stimulation are minimal. Accordingly, a reduction in cost-benefit by the use of wristband, is apparent. Considering the results from earlier research along with the promising results from our trial, we are encouraged to implement acupressure into our standard anaesthetic procedures. A reduction of the use of antiemetics will be a parameter on the effectiveness of acupressure.

The aim of this quality improvement study is to implement acupressure as a supplement to the ordinary prophylactic treatment of PONV in our hospital. The objective is to observe whether use of acupressure wristbands reduces the consumption of antiemetics for the treatment of postoperative nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Adults undergoing orthopaedic, general, and ear, nose, throat surgery at Lovisenberg Diaconal Hospital

Exclusion Criteria:

* Not fully verbal communication or informed consent not achieved

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2011-09; Primary Completion 2011-12 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of acupressure for postoperative nausea in terms of less use of antiemetic drugs | one year
  Study the effectiveness of acupressure for nausea in all surgical patients undergoing surgery at the Lovisenberg Diakonale hospital.
  Effectiveness is monitored by the use of antiemetic drugs compared to a similar period before the wristbands were introduced as standard care at the hospital.

SECONDARY OUTCOMES:
Reduction in use of antiemetic medication as a consequence of the introduction of acupressure wristband | One year
  The study will be conducted with a one-group pretest-posttest design, measuring the consumption of antiemetics during a three month period before the implementation (baseline), and during the implementation period. The numbers of surgical operations will be the denominator in the two fractions.
  This secondary outcome might also be regarded as the primary outcome as the amount of antinausea medication is the major outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Arne Johan Norheim, PhD, Principal Investigator — University of Tromso
Locations (1):
- Lovisenberg Diaconal Hospital, Oslo, Norway